CLINICAL TRIAL: NCT02124668
Title: A Phase 2, Multicenter, Single-arm, Open Label Study to Monitor the Safety of Enzalutamide in Patients With Progressive Castration-Resistant Prostate Cancer Previously Treated With Docetaxel-Based Chemotherapy
Brief Title: A Study to Monitor the Safety of Enzalutamide in Patients With Progressive Castration-Resistant Prostate Cancer Previously Treated With Docetaxel-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0122
Record Dates: First submitted 2014-04-25; First posted 2014-04-28 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Castration-Resistant Prostate Cancer; Prostate Cancer
Keywords: Xtandi; MDV3100; Progressive Castration-Resistant Prostate Cancer; Enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzalutamide (Experimental): Enzalutamide
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — oral
  Other Names: Xtandi; MDV3100

SUMMARY:
The purpose of this study is to monitor the safety of enzalutamide in patients with progressive castration-resistant prostate cancer previously treated with docetaxel-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically or cytologically confirmed adenocarcinoma of the prostate
* Subject has ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) analogue (agonist or antagonist) and plans to maintain throughout the study period or has had a prior orchiectomy (i.e., surgical or medical castration)
* Subject has had at least one prior chemotherapy regimen for metastatic castration-resistant prostate cancer with at least one regimen containing docetaxel
* Subject has progressive disease and indication for change of antineoplastic regimen
* Subject has no known or suspected brain metastasis
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Subject is able to swallow the study drug and comply with study requirements
* There is no comparable or satisfactory alternative therapy to treat the subject's disease
* Subject agrees not to participate in another interventional study while on treatment

Exclusion Criteria:

* Subject has severe concurrent disease, infection, or co-morbidity that would make the subject inappropriate for enrollment
* Subject's absolute neutrophil count is < 1000/μL, or platelet count < 100,000/μL, or hemoglobin < 6.2 mmol/L (or < 10 g/dL)
* Subject's total bilirubin is ≥ 1.5 x upper limit of normal (ULN) (except for subjects with documented Gilbert's disease) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is ≥ 2.5x ULN
* Subject's estimated creatinine clearance is less than 30 mL/min by the Cockcroft and Gault formula
* Subject has albumin ≤ 30 g/L (or ≤ 3.0 g/dL)
* Subject has received anti-androgen therapy (e.g. bicalutamide), chemotherapy, or biologic therapy for prostate cancer (other than bone targeted agents such as bisphosphonates or denosumab, gonadotropin-releasing hormone (GnRH) analogue therapy, or glucocorticoids which are allowed) within 4 weeks of Day 1
* Subject has had prior use of abiraterone
* Subject has prior use, or participation in a clinical trial, of an investigational agent that blocks androgen synthesis (e.g. TAK-700) or targets the androgen receptor (e.g. ARN-509, ODM-201)
* Subject has:

  1. A history of seizure, including any febrile seizure or any condition that may predispose to seizure including, but not limited to underlying brain injury, stroke, primary brain tumors, brain metastases,
  2. A history of loss of consciousness or transient ischemic attack within 12 months of Screening
* Subject has clinical signs suggestive of high or imminent risks for pathological fracture, spinal cord compression and/or cauda equina syndrome
* Subject has a significant cardiovascular disease
* Subject has received investigational therapy within 28 days or 5 half lives, whichever is longer, prior to Screening
* Subject has undergone major surgery within 4 weeks prior to Screening
* Subject has shown a hypersensitivity reaction to the active pharmaceutical ingredient or any of the capsule components, including Labrasol, butylated hydroxyanisole, and butylated hydroxytoluene
* Subject has used or plans to use, from 30 days prior to enrollment through the end of the study, medications known to lower the seizure threshold or prolong the QT interval

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Safety profile of enzalutamide assessed by adverse events (AEs), serious AEs (SAEs), vital signs, electrocardiograms (ECGs) and laboratory measurements | Up to 30 days after the last dose of enzalutamide or prior to the initiation of another anticancer therapy, whichever comes first (up to 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (4):
- Georgia (2):
  - Site GE99503, Tbilisi
  - Site GE99502, Tbilisi
- Russia (2):
  - Site RU70002, Moscow
  - Site RU70003, Moscow

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=250